CLINICAL TRIAL: NCT04638179
Title: Efficacy of Multi-disciplinary Integrated Post-acute Care in Patients Admission for Heart Failure
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006182RIND
Record Dates: First submitted 2020-10-30; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2018-02

CONDITIONS: Hospitalization Rate; Mortality Rate; Functional Recovery; Left Ventricle Ejection Fraction; NT-pro BNP
Keywords: National Health Insurance Administration post-acute care program; Heart Failure; multi-disciplinary integrated
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HF-PAC: (1) The experimental group is a patient who was managed by the NHIA 's acute post-care plan. Provide interdisciplinary comprehensive care in accordance with the norms and conduct health education during hospitalization. Hospitalized Chinese pharmacists, dietitians, physiotherapists and case managers participate in health education and will continue to be interviewed and have heart consultations within six months of discharge.
  Interventions: Other: Not intervention.Use retrospective case contrl study.
- HF-non PAC: (2)The control group received traditional health education in general care and routine health care.

INTERVENTIONS:
Other: Not intervention.Use retrospective case contrl study. — Use retrospective case contrl study.
  Other Names: Use retrospective case contrl study.
  Groups: HF-PAC

SUMMARY:
Background: Clinical heart failure patients always suffering from (1) worsen symptoms such as decreased activity tolerance, end-to-end breathing and excessive body fluid volume; (2) high medical expenses results from hospitalization; (3) reduced quality of life . In 2018, following instruction from National Health Insurance Administration (NHIA), the National Taiwan University Hospital (NTUH) undertook National Health Insurance post-acute care program, PAC in charge of heart failure patients by multi-disciplinary integrated to reduce acute exacerbations(AE), control symptoms, improve quality of life and increase survival rate.

DETAILED DESCRIPTION:
Objective: To evaluate the outcome of patients with heart failure who been taken are of multi-disciplinary integrated instructed by National Health Insurance Administration (NHIA)

Methods: Use retrospective case contrl study. Adopted the hospitalized patients diagnosed with heart failure in the NTUH as the research sample, and collected the retrospective data for analysis in a two-group study design. (1) The experimental group is a patient who was managed by the NHIA 's acute post-care plan. Provide interdisciplinary comprehensive care in accordance with the norms and conduct health education during hospitalization. Hospitalized Chinese pharmacists, dietitians, physiotherapists and case managers participate in health education and will continue to be interviewed and have heart consultations within six months of discharge. (2)The control group received traditional health education in general care and routine health care.

Time of review: From February 2, 2018, the implementation of the National Health Insurance Agency's acute post-care plan day to December 31, 2019, and continuous tracking of effectiveness for one year.

Exclusion conditions: (1) Age over20 years, (2) long-term dialysis, (3) unconsciousness, (4) complete bed rest without self-care ability, (5) those with ventilator dependence, (6) ventricular assist device (VAD) has been implanted, (7) heart transplants , (8) refused to join the research.

The monitoring indicators: Hospitalization rate within 180 days, mortality rate within one year , functional recovery, left ventricle ejection fraction (LVEF), NT-pro BNP, etc.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Heart Failure

* The experimental group is a patient who was managed by the NHIA 's acute post-care plan. Provide interdisciplinary comprehensive care in accordance with the norms and conduct health education during hospitalization. Hospitalized Chinese pharmacists, dietitians, physiotherapists and case managers participate in health education and will continue to be interviewed and have heart consultations within six months of discharge.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exclusion Criteria:
  * (1) Age over20 years, (2) long-term dialysis, (3) unconsciousness, (4) complete bed rest without self-care ability, (5) those with ventilator dependence, (6) ventricular assist device (VAD) has been implanted, (7) heart transplants , (8) refused to join the research.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Hospitalization rate within 180 days | within 180 days
  Hospitalization rate

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, No. 7, Zhongshan S. Rd., Zhongzheng Dist., Tai, Taiwan